CLINICAL TRIAL: NCT03631875
Title: Co-induction Ketamine-propofol: the Effects on Laryngeal Mask Airway Insertion Conditions and Resulting Hemodynamic Changes in Children
Brief Title: Co-induction Ketamine-propofol: Effects on Laryngeal Mask Airway Insertion Conditions in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Mahdia (Other)
Responsible Party: Principal Investigator, Majdoub Ali MD, head of anesthesia departement, University Hospital, Mahdia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Ketco1
Record Dates: First submitted 2018-07-02; First posted 2018-08-15 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Anesthesia Intubation Complication
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: After inhalatory induction with sevoflurane7%until abolition of the eye lash reflex, an intravenous canula was inserted in the dorsum of the hand. The sevoflurane concentration was then decreased to 2% in 100% O2.A nurse not involved in the study prepared two syringes with ketamine or normal saline, and administrated it according randomization , one minute before induction with propofol. The administration of propofol was realized on 60 seconds. An experimented anesthesiologist evaluated the LM conditions insertion. When the jaw was relaxed, and deglutition and cough reflex and member movement were absent, the conditions were considered acceptable. The LM was then inserted. For analgesia,we proceeded by a locoregional bloc adapted to the surgery. We recorded systolic and diastolic blood pressure, HR and SpO2 at the induction time at LM insertion and at the 3rd,5th and10th min.
Who Masked: Outcomes Assessor
Masking Description: A nurse not involved in the study prepared two syringes with ketamine or normal saline, and administrated it according randomization (by computer generated random numbers) one minute before induction with propofol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P (propofol), (Placebo Comparator): normal saline is injected 01 min before induction with propofol 3 mg/kg. After 60 seconds, an experimented anesthesiologist evaluated the LM conditions insertion.
  Interventions: Drug: Ketamine
- PK (propofol-ketamine) (Active Comparator): we inject 0.5 mg/kg of ketamine 01 min before induction with 03 mg/kg of propofol .Sixty seconds after, an experimented anesthesiologist evaluated the LM conditions insertion.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — use a low dose 0.5 mg/kg of ketamine in coinduction with propofol in children induction anesthesia
  Other Names: co-induction ketamine propofol

SUMMARY:
Background: Large doses of propofol needed for induction and laryngeal mask (LM) insertion in children may be associated with hemodynamic sides effects. Co-induction with low doses of ketamine 0.5 mg/ kg has the advantage of reducing dose and therefore maintaining hemodynamic stability.

Aim: To examine the effect of co-induction on LM insertion, hemodynamics and recovery in children

DETAILED DESCRIPTION:
A prospective, randomized, double-blind, controlled study was conducted including120 ASA physical status I ⁄ II unpremedicated children, aged 1-8 years. Inhalatory induction with sevoflurane at 7% to insert an intravenous canula was first used then decreased to 2%. Normal saline or ketamine (0.5 mg/kg) were administered in groups P (propofol), PK (propofol-ketamine) respectively, 1 min prior to the administration of the induction dose of propofol. Propofol 3mg/kg was used for induction in the 2 groups, LM inserted 60 s later and insertion conditions assessed. Heart rate and blood pressure were recorded immediately after propofol bolus, then after LM insertion, at the 3rd ,5th and 10th minutes later. Recovery was assessed using Steward's Score

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status I and II
* unpremedicated
* ambulatory surgery

Exclusion Criteria:

* surgery complication
* upper air way complications

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
laryngeal masque conditions insertion | MINUTE 1
  When the jaw was relaxed, and deglutition and cough reflex and member movement were absent, the conditions were considered acceptable.the laryngeal masque was inserted

SECONDARY OUTCOMES:
hemodynamic conditions | HOURS 1
  systolic blood pressure
heart rate | HOURS 1
  cardiac frequence

CONTACTS AND LOCATIONS:
Overall Officials: ali majdoub, professor, Study Director — Ministery of Health
Locations (1):
- Mahdia University Hospital, Mahdia, Tunisia

IPD SHARING:
Plan to Share IPD: No